CLINICAL TRIAL: NCT04887298
Title: Phase 1B/2 Study of Liposomal Annamycin (L-Annamycin) in Subjects with Previously Treated Soft-Tissue Sarcomas with Pulmonary Metastases
Brief Title: Study of Liposomal Annamycin for the Treatment of Subjects with Soft-Tissue Sarcomas (STS) with Pulmonary Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Moleculin Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MB-107
Record Dates: First submitted 2021-05-04; First posted 2021-05-14 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Sarcoma,Soft Tissue; Pulmonary Metastasis
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liposomal Annamycin (L-Annamycin) (Experimental)
  Interventions: Drug: Liposomal Annamycin (L-Annamycin)

INTERVENTIONS:
Drug: Liposomal Annamycin (L-Annamycin) — 2-hour intravenous (IV) infusion of L-Annamycin on Day 1 followed by 20 days off of study drug (i.e., 1 treatment cycle= 21 days)

SUMMARY:
This is a multi-center, open-label, single-arm study that in Phase 1b will determine the maximum tolerated dose (MTD)/ recommended phase 2 dose (RP2D) and safety of L-Annamycin and in Phase 2 will explore the efficacy of L- Annamycin as a single agent for the treatment of subjects with STS with lung metastases for which chemotherapy is considered appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a pathologically confirmed diagnosis of STS.
2. The subject must have radiographically measurable disease in the lung that can be assessed using RECIST v.1.1 (defined as the presence of at least one lesion on MRI or CT scan that can be accurately measured with the longest diameter in at least one dimension of ≥10 mm). Subjects with extra-pulmonary disease are eligible.
3. The subject has documented lung metastases that are considerable eligible for chemotherapy and not eligible for potentially curative surgical resection of pulmonary-only metastatic disease.
4. The subject had prior therapy for their disease and has shown progression of disease prior to study entry. If the subject received prior anthracycline therapy, they must have received a cumulative dose of ≤ 450 mg/m2.
5. The subject has an estimated life expectancy of greater than 3 months.
6. The subject has an ECOG performance status ≤2.
7. The subject is ≥18 years old at the time of signing informed consent.
8. At least 2 weeks must have passed following treatment for subject's disease with chemotherapy, investigational therapy, targeted agents, biological agents, immune modulators, or radiotherapy.
9. Any toxicities must have resolved to ≤ grade 1 or previous baseline levels no more than 4 weeks after completing therapy (except alopecia and polyneuropathy).
10. The subject must have the following adequate laboratory results within 72 hours of starting protocol therapy:

    1. Absolute neutrophil count ≥ 1500/mL
    2. Platelet count ≥100,000/mL
    3. Hemoglobin ≥ 8.0 g/dL
    4. Adequate renal function (The Cockcroft-Gault equation will be used to estimate creatinine clearance.

       CrCl (male) = ([140-age] x weight in kg) / (serum creatinine x 72)

       CrCl (female) = ([140-age] x weight in kg) / (serum creatinine x 72) x .85
    5. Bilirubin ≤1.5 x ULN (unless due to Gilbert's syndrome)
    6. Aspartate aminotransferase (serum glutamic oxaloacetic transaminase) and/or alanine aminotransferase (serum glutamic pyruvic transaminase) ≤ 2.5 × ULN (≤ 5 x ULN in subjects with liver metastases)
11. The subject is able to understand and sign the informed consent document, can communicate with the Investigator, and can understand and comply with the requirements of the protocol.
12. All subjects must agree to practice effective contraception during the entire study period and after discontinuing study drug, unless documentation of infertility exists.

    1. Sexually active, fertile women must agree to use 2 effective forms of contraception (abstinence, intrauterine device, oral contraceptive, or double barrier device) from the time of informed consent and until at least 6 months after discontinuing study drug
    2. Sexually active men and their sexual partners must agree to use effective contraceptive methods from the time of informed consent until at least 6 months after discontinuing study drug

Exclusion Criteria:

1. The subject has any uncontrolled intercurrent illness that, in the opinion of the Investigator, would place the subject at unacceptable risk to participate in the study. Examples include, but are not limited to:

   1. Ongoing or active infection
   2. Known positive status for human immunodeficiency virus (HIV) or active hepatitis B or C
   3. Cirrhosis
   4. Psychiatric illness/social situations that would limit compliance with study requirements
2. The subject has any of the following cardiotoxicities:

   1. Left ventricular ejection fraction (LVEF) <50%
   2. Valvular heart disease
   3. Severe hypertension not controlled by medical therapy
   4. New York Heart Association classification of 3 or 4 (Appendix B)
   5. Recent (≤ 6 months) myocardial infarction
   6. Unstable angina
   7. Symptomatic congestive heart failure
   8. Baseline QT/QTc interval >480 msec
   9. History of additional risk factors for torsade des pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
   10. Use of concomitant medications that significantly prolong the QT/QTc interval
3. The subject is pregnant (must have negative serum or urine pregnancy test) or lactating.
4. The subject has a known allergy to study drug, L-Annamycin, or excipients.
5. The subject is required to use moderate or strong inhibitors and inducers of Cytochrome P450 family enzymes CYP3A and CYP2B and transporters that cannot be held 3 days before treatment and on the day of treatment (Appendix E).
6. The subject is unable to comply with the safety monitoring requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 21 days
  Number of patients with a dose limiting toxicity (DLT) at each dose evaluated

SECONDARY OUTCOMES:
Efficacy of L-Annamycin | At the end of every other treatment cycle ( each cycle is 21 days)
  Determine preliminary efficacy of L-Annamycin as per revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1)
Area Under the Plasma Concentration Versus Time Curve (AUC) of L-Annamycin | Cycle 1 Day 1 ( each cycle is 21 days)
  Determine pharmacokinetics of L-Annamycin and its metabolite, annamycinol as measured by AUC

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shepard, MD, Study Director — Moleculin Biotech, Inc.
Locations (5):
- United States (5):
  - Sarcoma Oncology Center, Santa Monica, California
  - Washington University, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No